CLINICAL TRIAL: NCT03099733
Title: Development and Implementation of a Real-Time Assessment and Intervention for mTBI Patients Post-Discharge From the Emergency Department
Brief Title: Concussion Texting Study
Acronym: texting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 07-16-04A
Record Dates: First submitted 2017-02-06; First posted 2017-04-04 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2019-03

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- concussion (Experimental): patients who present to ED with concussion
  Interventions: Other: text message

INTERVENTIONS:
Other: text message — Participants will receive text message assessment and tailored intervention messages daily over the 14-day/two-week study period.

SUMMARY:
This will be a prospective study of the implementation of a real-time assessment and intervention of a text messaging tool in mild traumatic brain injury (mTBI) patients post-discharge from the emergency department.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is an important cause of morbidity and mortality in children, resulting in an estimated 173,000 emergency department (ED) visits and 14,000 hospitalizations each year in the US. The estimated rate of TBI visits increased 57% from 2001-2009, and in 2010 there were more than 2.5 million TBI-related ED visits. Most patients are discharged from the ED and diagnosed with a closed head injury, minor head injury, concussion, or other unspecified head injury. After discharge, patients, family members, and other care partners may report certain mTBI symptoms that may lead to unnecessary utilization of healthcare services.

Novel, effective, and cost-effective solutions for mTBI symptom management post ED discharge are needed to improve the patient's understanding about their symptoms after discharge. Use of mobile technology to interact with mTBI patients may: 1) extend the reach of clinicians, 2) offer patients diagnosed with a mTBI a form of ongoing tailored clinical support, and 3) contribute to improved health outcomes and optimization of health care utilization. Previous research shows high compliance with text-message based interventions, measurable change in behavior, and prolonged adherence to clinical guidance. A recent randomized trial of mTBI patients showed high-compliance with text-message assessments following ED discharge, and a trend towards fewer and less severe post-mTBI symptoms in the intervention group. The investigators propose to develop and pilot a novel mobile phone text-messaging platform to perform real-time assessment and intervention of mTBI patients discharged from the ED. This intervention will empower patients to actively participate in the management of their condition. Use of this technology with the mTBI patient population is feasible and cost-effective. Over 90% of Americans own a cell phone or smartphone, and 80% send and receive text-messages.

The first objective of this research study is to develop and pilot the novel use of an existing technology, mobile phone text-messaging, to perform real-time assessment and feedback regarding symptoms of mTBI patients post-discharge from the ED. A second objective is to assess the effect of a brief, real-time, tailored intervention designed to impact patient and caregiver understanding of their mTBI related symptoms. The overarching goal of this proposal is to build on the work of Dr. Hirsch, et al. who found that: 1) mTBI patients report a poor understanding of concussion; 2) mTBI patients reported insufficient communication with clinicians regarding their symptoms following ED discharge (e.g., balance and sleep); and 3) mTBI patients reported poor care coordination, poor follow-up, and limited access to specialist physicians post-discharge.

Hypothesis: Based on prior work, implementation of a text-based tool for assessment and intervention of mTBI patients post-discharge from the CMC-Main & LCH EDs will improve patient engagement related to mTBI. It is anticipated that 50% of potential study subjects will elect to receive text messages and that the differences in characteristics of enrolled participants versus non-participants will not be statistically significant. It is anticipated that > 75% of participants will respond/comply with the symptom assessment messages.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or greater and diagnosed with a concussion or closed head injury with intent to discharge from the ED
* Blunt trauma mechanism of injury
* GCS 14 or greater upon arrival to the ED
* The patient or caregiver owns a cell phone with text messaging capability

Exclusion Criteria:

* Penetrating trauma mechanism of injury
* The patient or caregiver does not own a cell phone with text messaging capability or is unwilling to receive text messages
* If the patient has a condition that makes him/her unable to communicate via text message
* Known unavailability (travel, planned surgery, etc.) during the follow-up period
* Planned admission to the hospital
* Abnormal CT, if obtained
* Social issues that preclude follow-up
* Alcoholism
* Major psychiatric or personality disorder
* Incarceration or arrest
* Baseline cognitive impairment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | Study duration (one year, anticipated)
  The intervention will be determined to be feasible if the majority of subjects respond to the text messages and complete follow-up, and if the majority of subjects that are approached agree to participate. The demographic and baseline characteristics of participants and non-participants will be assessed for significant differences that may have influenced the feasibility assessment.

SECONDARY OUTCOMES:
Identify obstacles associated with the text messaging instrument | 14 days
  Qualitative interview with participants by phone - participants will be asked about their thought and feelings related to the study assessment tool, relationships with the study physicians, text messaging impact on care and recommended changes.
Healthcare utilization | 3 months
  To gauge the safety and effectiveness of the intervention, we will determine if there are patient level factors that increase the rate of follow-up and decrease direct cost of care.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Scarboro, MD, Principal Investigator — Carolinas Medical Center/Atrium Health
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No